CLINICAL TRIAL: NCT00334347
Title: A Comparison Study of the Efficacy and Tolerability Between Depakote ER and Depakote in the Acute Treatment of Mania and Mixed Mania
Brief Title: A Comparison Study of the Efficacy and Tolerability of Depakote ER and Depakote DR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: John D. Matthews, MD, Massachusetts General Hospital, Boston, Massachusetts 02114
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-P-000671
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-12

CONDITIONS: Mania; Mixed Mania
MeSH Terms: conditions — Mania | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depakote ER (Active Comparator)
  Interventions: Drug: Depakote ER
- Depakote DR (Active Comparator)
  Interventions: Drug: Depakote DR

INTERVENTIONS:
Drug: Depakote ER — The starting doses will be 25 mg/kg and 20 mg/kg. The dose you get will depend on how much you weigh.
  Arms: Depakote ER
Drug: Depakote DR — The starting doses will be 25 mg/kg and 20 mg/kg. The dose you get will depend on how much you weigh.
  Arms: Depakote DR

SUMMARY:
To compare the time to response, response rates, remission rates, and side effects in Bipolar Disorder inpatients treated with Depakote ER or Depakote DR for acute mania or mixed mania.

DETAILED DESCRIPTION:
There are several studies demonstrating the efficacy of divalproex in the acute treatment of mania and mixed mania. In fact, the American Psychiatric Associations Practice Guidelines for Bipolar Disorder recommends divalproex as a first-line treatment for acute mania and acute mixed mania; divalproex is the treatment of choice in the treatment of acute mixed mania. The Food and Drug Administration (FDA) approved divalproex for the acute treatment of mania in the 1990's. A new formulation, divalproex, Depakote ER, was recently FDA approved for the treatment of epilepsy and prophylaxis of migraine headaches. In a pooled data analysis of nine open-labeled trials involving 321 epilepsy and bipolar disorder patients, Smith et al. that Depakote ER was associated with superior tolerability including less frequent tremors, weight gain, and gastrointestinal complaints (all p<0.001) compared with Depakote DR. Depakote ER was preferred by subjects and it provided improved seizure control and a greater reduction in psychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages 19-65 (inclusive).
* DSM-IV diagnosis of acute mania or acute mixed mania .

Exclusion Criteria:

* DSM-IV diagnoses of bipolar disorder, depressed type, bipolar disorder rapid cycling type, major depressive disorder with psychotic features, schizoaffective disorder, schizophrenia, substance use disorder (active use within the last 3 months), or organic mood disorder.
* History of a seizure disorder or an unstable physical disorder judged to significantly affect central nervous system function.
* Female subjects who are pregnant or of childbearing potential who are not using medically accepted means of contraception and female patients who are breastfeeding.
* Subjects who require antipsychotic medications because of severe psychosis and /or agitation.
* Subjects on antidepressants or mood stabilizers including lithium, oxcarbazepine, carbamazepine, and lamotrigine.
* Subjects who have failed previous trials with Depakote DR or Depakote ER.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The Young Mania Rating Scale (YMRS)will be used daily for the first week and then every three day to assess the severity of mania. | study duration
The Clinical Global Impression Scale (CGI) will be used daily for teh first week then every 3 days to assess overall functioning. | study duration
The Udvalg for Kliniske Undersogeiser (UKU) Side Effect Rating Scale will be administered at base line and weekly for the remainder of the study to determine the medication side effect profiles. | study duration

SECONDARY OUTCOMES:
The Montgomery-Asberg Depression Rating Scale will be performed daily for the first week and weekly thereafter to assess for any emergent symptoms of depression. | study duration
The Brief Psychiatric Rating Scale (BPRS) will be performed daily for the first week and weekly thereafter to assess for any emergent symptoms of psychosis. | study duration
The Drug Attitude Inventory (DAI-10)will measure subjects' attitudes towards medications at the screen and final visit. | study duration
The Schizophrenia Quality of Life Scale (SQLS)will measure subjects' quality of life at the screen and final visit. | study duration

CONTACTS AND LOCATIONS:
Overall Officials: John D Matthews, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States